CLINICAL TRIAL: NCT02362191
Title: Targeting Inter-Hemispheric Alpha Coherence With tACS To Treat PMDD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated because the dense treatment schedule precluded successful recruitment of study participants.
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Foundation of Hope, North Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-0600
Record Dates: First submitted 2014-09-27; First posted 2015-02-12 (Estimated); Results first posted 2020-10-09 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-06

CONDITIONS: Premenstrual Dysphoric Disorder
MeSH Terms: conditions — Premenstrual Dysphoric Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Session tACS Across Menstrual Cycle (Experimental): Participants assigned to receive a single session of tACS during the follicular and luteal phase of their menstrual cycle.
  Interventions: Device: Alternating Current Stimulator

INTERVENTIONS:
Device: Alternating Current Stimulator — Transcranial alternating current stimulation (tACS) is a method of noninvasive brain stimulation in which weak electrical current are applied to the scalp in a sine wave pattern to induce cortical oscillations at the frequency at which they are applied.
  Other Names: XCSITE 100 Stimulator

SUMMARY:
Purpose: Using transcranial alternating current stimulation (tACS), we will study whether tACS induces changes in prefrontal alpha oscillatory frequencies in women with premenstrual dysphoric disorder (PMDD) and whether tACS effects on alpha oscillations varies by menstrual cycle phase. An exploratory objective is to assess whether there are any changes in symptom severity during the menstrual cycle phase in which tACS is delivered relative to their baseline symptom levels (determined in a diagnostic feeder study, see below).

Participants: Women between ages 18-52 with a diagnosis of PMDD confirmed by participation in a PMDD diagnostic study (IRB# 05-3000).

Procedures (methods): After a re-screening and consent appointment, eligible participants will alert the study staff when they begin menstruating. Participants will have their first session in either the follicular phase or luteal phase (determined by ovulation testing) of their menstrual cycle and the second session in the other cycle phase. The order of phase at first testing will be counterbalanced across participants. Each session will consist of 40 minutes of tACS with by an EEG recording before and after stimulation. Patients' symptoms will be assessed at the end of each session and with the daily mood ratings collected throughout the menstrual cycle that coincides with tACS sessions (approximately 26 - 32 days).

DETAILED DESCRIPTION:
Premenstrual Dysphoric Disorder (PMDD) describes the cyclic appearance of affective symptoms and resultant impairment during the luteal phase of the menstrual cycle. The objective of the experiment is to determine if transcranial alternating current electrical stimulation (tACS) will alter prefrontal alpha oscillatory frequencies in women with PMDD, disruption of which has been implicated in other mood disorders. A secondary objective is to determine if menstrual cycle phase will influence the effects of tACS on alpha oscillations. Demonstration of 'target engagement' (alterations in left prefrontal alpha oscillatory frequencies with tACS) is a necessary first step before moving forward with subsequent research that would test whether tACS is a potential treatment for this disorder - promising research in other mood disorders suggests that it may be.

The cause of PMDD is unknown, the morbidity substantial, and the identified treatments limited in their effectiveness, since 40% of PMDD women are non-responders to SSRIs and many additional women are intolerant of antidepressant induced side effects. PMDD is prevalent (6-8% of women of reproductive age), attended by substantial morbidity, and hence a significant public health problem. Indeed, by World Health Calculations, PMDD is associated with 4.5 million Disability Adjusted Life Years in the US alone. The rationale for testing whether tACS differentially alters target engagement in the follicular versus luteal phases of the menstrual cycle is described below.

Differential Effects on Cortical Activity: The rationale for testing whether tACS differentially alters target engagement in the follicular versus luteal phases of the menstrual cycle is as follows: 1) Role of Hormones: While there is little evidence for ovarian dysfunction in PMDD a role for the reproductive hormones is clearly implicated, since our own work and that of others has shown that suppression of ovarian function results in a complete remission of symptoms in a majority of women with PMDD, while adding back gonadal hormones results in the return of symptoms in women with PMDD, with no symptoms seen in controls. Both estradiol and progesterone appear capable of precipitating mood destabilization in this paradigm. Recently completed studies from our group further demonstrate that continuous administration of hormones for longer than one-month results in a sustained symptom remission subsequent to the initial precipitated episode. Thus, dysphoric mood states in PMDD appear to be induced by normal changes in gonadal hormones rather than by exposure to elevated hormone levels (i.e., women with PMDD are differentially sensitive to the mood dysregulatory effects of reproductive steroids).

Although there is substantial literature demonstrating the effects of reproductive steroids and, by extension, the menstrual cycle on cortical activity, the usually described effects are disturbed in women with PMDD. Examples include the following: 1) in normal women, activation of the medial orbitofrontal cortex is diminished during the luteal phase and the affective valence of the stimulus to which it responds is reversed (i.e., it responds only to negative stimuli rather than to positive stimuli, as occurs during the follicular phase). These changes are absent in women with PMDD. 2) in normal women during the luteal phase, there is an increase in cortical inhibition - a presumed effect of the GABA receptor activating effects of the progesterone metabolite allopregnanolone. This effect is absent in women with PMDD. Both animal and human data further suggest the role of a disturbed cortical response to progesterone-derived neurosteroids in PMDD. Thus, sudden changes in the levels of allopregnanolone (as occurs at the start of the luteal phase with increasing levels of progesterone) result in subcortical excitability and irritability in rodents, while elimination of changes in progesterone-derived neurosteroids (with neurosteroid synthesis inhibition) successfully prevents the emergence of the dysphoric state in PMDD.

Differential Network Activation: Psychiatric disorders characterized by dysregulation of affective state -depression and PMDD - are increasingly recognized as are "network disorders" in which aberrant electric signaling in large-scale neuronal networks mediates the clinical symptoms. Recent studies have documented impaired balance in activation between left and right prefrontal cortex in patients with PMDD. In particular, similar to major depressive disorder, the balance between alpha oscillation power in the left and the right hemisphere is shifted towards the left in patients with PMDD. The presence of alpha oscillations corresponds to a relative decrease in neuronal activity (inverse relationship). Therefore, such a left-shifted alpha asymmetry is indicative of hypoactivation of the left hemisphere - a common finding in imaging studies of patients with MDD. Since this asymmetry is exacerbated during the luteal but not the follicular phase (corresponding to the time course of symptom presentation in PMDD, we hypothesize that successful normalization of alpha oscillations in women with PMDD would be a plausible approach to symptom remediation. This network level intervention can be accomplished with brain stimulation by application of weak electric currents, a non-invasive approach to modulating intrinsic cortical network dynamics. The advantage of this approach is twofold: it is non-pharmacologic and thus avoids the otherwise attendant side effects; and it will provide systems level insights into the pathophysiology underlying mood state dysregulation.

Brain stimulation by constant electric currents applied to the scalp (tDCs) modulates neuronal excitability in humans. Transcranial current stimulation with sine-wave stimulation waveforms (transcranial alternating current stimulation, tACS) likely enhances cortical oscillations in a frequency specific manner. The mechanisms of weak electric fields generated by tDCS and tACS previously have been demonstrated to interact with cortical network activity by altering the temporal activity structure of electric signaling in cortex. In this study, we will assess whether tACS will decrease left frontal alpha power (8-12 Hz) and whether the extent of the decrease varies by menstrual cycle phase. An exploratory objective will be to examine the severity of the PMDD symptoms collected daily during the stimulation cycle and compare that severity with baseline symptoms ratings collected during the PMDD diagnostic study from which these participants will be recruited. The rationale for this stimulation is the known deficits in the overall structure of cortical activity in this frequency band in patients with mood disorders and the previously demonstrate clinical benefits of tDCS in the treatment of mood disorders. In this study, we will use more targeted stimulation waveforms by employing bilateral tACS instead of tDCS. We hypothesize that this choice of a more sophisticated waveform that directly enhances synchronization between the two hemispheres may be more effective in engaging the target. tDCS modulates overall activity levels of the targeted cortical area in a non-specific manner. Here, however, we propose to evaluate a more specific stimulation modality, tACS, (10 Hz stimulation frequency) that has been shown to selectively enhance cortical alpha rhythms. Since the selected patient population reportedly exhibits specific deficits in the alpha frequency band, our stimulation approach will provide a more targeted and therefore possibly a more effective manipulation.

Protocol History: This protocol was originally designed to test the therapeutic efficacy of tACS in PMDD in a double blind, randomized, sham controlled, cross-over study of 5 tACS sessions. We were unable to recruit subjects, largely consequent to the many daily treatment sessions required. We subsequently changed the primary focus of the study to that of determining whether a single session of tACS engaged left prefrontal cortical alpha oscillations and, by reducing them, reduced alpha asymmetry. We further asked whether this effect was menstrual cycle phase-dependent.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-52;
* Have participated in our PMDD diagnostic study (IRB# 05-3000);
* Regularly menstruating without hormonal contraceptives (e.g., birth control pills, injections, implants, progestin IUDs);
* Medication free or regularly taking medication that has no effect on the nervous system;
* Not currently pregnant or planning to become pregnant;
* With sufficient resources to prevent pregnancy

Exclusion Criteria included:

* Brain surgery or brain implants, including cochlear implants or aneurysm clips
* Neurological disease, like epilepsy or a brain tumor
* Traumatic brain injury
* Pregnant or nursing
* An unstable medical illness, like congestive heart failure or end stage kidney disease
* History of severe or recurrent substance abuse, or any substance abuse within 2 years of study enrollment
* History of suicidal behavior within 5 years of study enrollment

  * Department of Psychiatry Faculty, Employee, or Trainee

Ages: 18 Years to 52 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2015-03; Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R Rubinow, MD, Principal Investigator — Dept of Psychiatry, UNC School of Medicine

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Session tACS Across Menstrual Cycle
Started | 5
Completed | 3
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Single Session tACS Across Menstrual Cycle
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.8 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Alpha Frequency Electrical Activity in Left Frontal Cortex Following Stimulation
Description: Fast Fourier transform is applied to 8 minutes of EEG data before and after tACS. Primary outcome is the difference in alpha frequency amplitude (8-12 Hz) in the left frontal cortex from baseline as a result of intervention.
Time Frame: 8-minute recording before vs after intervention
Measure: Mean (Standard Deviation); unit: microvolts
Arm/Group | Single Session tACS Across Menstrual Cycle
Number analyzed (Participants) | 3
microvolts | 0.044 (0.218)
Statistical Analysis 1: Comparison: Single Session tACS Across Menstrual Cycle; Test type: Other; p = 0.758, t-test, 2 sided — The threshold for statistical significance is 0.05

2. Secondary Outcome: Difference in Magnitude of Effect of tACS on Left Prefrontal Alpha in Follicular vs Luteal Phase
Description: Comparison of the change in EEG left prefrontal activity following tACS in luteal vs. follicular phases measured by the luteal pre to post change in EEG compared with the follicular pre to post change in EEG. Pre-post EEG recordings will occur during the follicular phase (5-9 days after menstruation) and in the luteal, premenstrual phase (9-13 days after ovulation).
Time Frame: Over the course of 2 menstrual cycles, pre-post EEG recordings will occur, one during the follicular phase (5-9 days after menstruation) and one in the luteal, premenstrual phase (9-13 days after ovulation)
Measure: Mean (Standard Deviation); unit: microvolts
Arm/Group | Single Session tACS Across Menstrual Cycle
Number analyzed (Participants) | 3
microvolts | -0.191 (0.313)
Statistical Analysis 1: Comparison: Single Session tACS Across Menstrual Cycle; Test type: Other; p = 0.40, t-test, 2 sided — The threshold for statistical significance is 0.05

ADVERSE EVENTS:
Time Frame: Adverse events were collected starting at Baseline through the onset of menses after the second tACS session, an approximate total duration of up to 2 months
Arm/Group | Single Session tACS Across Menstrual Cycle
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-14): https://cdn.clinicaltrials.gov/large-docs/91/NCT02362191/Prot_SAP_000.pdf